CLINICAL TRIAL: NCT04162353
Title: BCMA-CD19 cCAR in Relapsed and /or Refractory Multiple Myeloma and Plasmacytoid Lymphoma
Brief Title: BCMA-CD19 cCAR in Multiple Myeloma and Plasmacytoid Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: iCAR Bio Therapeutics Ltd. (Industry); Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICG185-001
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma in Relapse; Refractory Multiple Myeloma; Plasmacytoid; Lymphoma
Keywords: BCMA; CD19; BCMA-CD19 cCAR T cells; multiple myeloma; plasmacytoid lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma

STUDY DESIGN:
Intervention Model Description: Dose escalation phase: BCMA-CD19 cCAR T cells transduced with a lentiviral vector to express two distinct units of BCMA and CD19 CARs on a T cell with an escalation approach, 2e6 to 10e6 CAR-T cells/kg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCMA-CD19 cCAR (Experimental): Dose escalation phase: BCMA-CD19 cCAR T cells transduced with a lentiviral vector to express two distinct units of BCMA and CD19 CARs on a T cell with an escalation approach, 2e6 to 10e6 CAR-T cells/kg
  Interventions: Biological: BCMA-CD19 cCAR T cells

INTERVENTIONS:
Biological: BCMA-CD19 cCAR T cells — BCMA-CD19 cCAR T cells administered to patients, will be either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of BCMA-CD19 cCAR in patients with relapsed and/or refractory multiple myeloma and plasmacytoid lymphoma.

DETAILED DESCRIPTION:
BCMA-CD19 cCAR is a compound Chimeric Antigen Receptor (cCAR) immunotherapy with two distinct functional CAR molecules expressing on a T-cell, directed against the surface proteins BCMA and CD19. BCMA-CD19 cCAR is also aimed to treat multiple myeloma, a challenging disease due to the heterogeneity of myeloma cells, which renders single-antigen targeting CAR T-cell therapy ineffective. BCMA-CD19 cCAR is proposed to target both bulky myeloma cells expressing BCMA, and myeloma stem cells expressing CD19 to effectively eradicate the disease.

BCMA-CD19 cCAR is also aimed to treat heterogeneous plasmacytoid lymphoma bearing two types of lymphoma cells, regular lymphoma cells expressing CD19 and plasmacytoid lymphoma cells expressing BCMA. The use of two different targets intends to increase coverage and eradicate cancerous cells before resistance develops in surviving cancer cells that have undergone selective pressures or antigen escape.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent; Patients volunteer to participate in the research
* Diagnosis is mainly based on the World Health Organization (WHO) 2008
* Patients have exhausted standard therapeutic options
* Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 1 weeks
* Female must be not pregnant during the study

Exclusion Criteria:

* Patients declining to consent for treatment
* Prior solid organ transplantation
* Potentially curative therapy including chemotherapy or hematopoietic cell transplant
* Prior treatment with BCMAxCD3 or CD19xCD3 bispecific agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events after BCMA-CD19 cCAR T cells infusion | 2 years particularly the first 28 days after infusion
  Determine the toxicity profile of BCMA-CD19 cCAR T cell therapy

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | up to 6 months
  Incidence of treatment-emergent adverse events

OTHER OUTCOMES:
For multiple myeloma - Stringent complete response | 24 months
  Stringent complete response (sCR) (IMWG criteria)
For multiple myeloma - Complete response (CR) | 24 months
  Complete response (CR) (IMWG criteria)
For multiple myeloma - Very good partial response (VGPR) | 24 months
  Very good partial response (VGPR) (IMWG criteria)
For multiple myeloma - Partial response (PR) | 24 months
  Partial response (PR) (IMWG criteria)
For multiple myeloma - Minimal response (MR) | 24 months
  Minimal response (MR) (IMWG criteria)
For multiple myeloma - Stable disease (SD) | 24 months
  Stable disease (SD) (IMWG criteria)
For multiple myeloma - Progressive disease (PD) | 12 months
  Progressive disease (PD) (IMWG criteria)
For multiple myeloma - Progression-free survival (PFS) | up to 24 months
  Progression-free survival (PFS) (IMWG criteria)
For plasmacytoid lymphoma - Assessment of morphologic CR, CR1, no residual disease, and molecular remission | 1 year
  Assessment of morphologic complete remission (CR), complete remission with incomplete recovery of counts (CR1), no residual disease as analyzed by flow cytometry analysis, and molecular remission by molecular studies
For plasmacytoid lymphoma - Progression-free survival (PFS) | 1 year
  Progression-free survival (PFS)
For plasmacytoid lymphoma - Overall survival | 1 year
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhang, MD/PhD, Principal Investigator — Peking University Shenzhen Hospital, China; Fang Liu, MD/PhD, Principal Investigator — Chengdu Military General Hospital
Locations (2):
- China (2):
  - Peking University Shenzhen Hospital, China, Shenzhen, Guangdong
  - Chengdu Military General Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No